CLINICAL TRIAL: NCT05725733
Title: The Effect of Physical Activity on The Response of Autonomic Nervous System in Individuals With Autism Spectrum Disorders of Different Age Groups
Brief Title: The Effect of Physical Activity Autonomic Response of Autism Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Mohammed Moustafa, Assistant Professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2265749561
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A single- blinded randomized controlled study design will be used, the exercise program will be administrated for four weeks, three times per week, and sixteen minutes per session. Heart rate, ECG, Measurements of respiration, and blood pressure will be measured three times every session: at rest before starting exercises (baseline), directly after finishing exercises, and 15 minutes after finishing exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- children with ASD group. (Experimental): ASD groups will be randomly divided into 4 subgroups according to their age (4-7 years old, 7-10 years old, 10-13 years old and, 14-18 years old). Also, ASD group will be categorized according to the symptoms severity using the childhood autism rating scale (CARS).
  Interventions: Other: Physical Therapy
- One hundred typically developed children or control group (Active Comparator): They will be randomly divided into 4 subgroups according to their age (4-7 years old, 7-10 years old, 10-13 years old and, 14-18 years old)
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — The participant will walk for 3-minutes at this speed as a warming up period. After these 3-minutes, the speed will be increased gradually up to 5-6 km/minute under the supervision of parents and therapist. The children will perform 10-minute running at this speed. After this, the cooling down exercise will be performed for 3-minutes. The speed will be decreased for 2 km/ minute and gradually stop.
  Other Names: Treadmill walking program

SUMMARY:
This study will investigate the effect of physical activity on autism spectrum disorder (ASD) in individuals with ASD of different age groups through measuring the hemodynamic, heart activity and respiratory system parameters.

DETAILED DESCRIPTION:
One hundred participants will be included in this study. One hundred typically developed children or control group and one hundred children with ASD group. The age range of participants will be 4 - 18 years old. The participants in both control and ASD groups will be randomly divided into 4 subgroups according to their age (4-7 years old, 7-10 years old, 10-13 years old and, 14-18 years old). Also, ASD group will be categorized according to the symptoms severity using the childhood autism rating scale (CARS). Participants will be excluded if they have any intellectual disability (IQ ≤ 70), co-morbid medical or psychiatric disorders, pervasive developmental disorders (PDD) or Attention-deficit hyperactivity disorders (ADHD). They will also be excluded if they are taking any medications which to affect cardiovascular system, respiratory system, or arousal and balance or any other contraindications to exercises. Wechsler Intelligence Scale for Children-Fourth Edition24 will be used to assess the Intelligence Quotient (IQ).

ELIGIBILITY:
Inclusion Criteria:

1. Children with ASD group with the age range of participants will be 4 - 18 years old
2. Typically developed children with the age range of participants will be 4 - 18 years old

Exclusion Criteria:

Participants will be excluded if they have the following:

* any intellectual disability (IQ ≤ 70)
* co-morbid medical or psychiatric disorders.
* pervasive developmental disorders (PDD) or Attention-deficit hyperactivity disorders (ADHD).
* They will also be excluded if they are taking any medications which to affect cardiovascular system, respiratory system, or arousal and balance or any other contraindications to exercises.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
ECG measurements | One minute
  A wearable device will be used to collet cardiac ECG data.
Measurements of respiration | 5 minutes
  Portable Respiratory Monitor will be used to measure the respiratory activity.
Blood pressure measurement | 5 minutes
  Manual sphygmomanometer will be used to measure the blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Ahmed, Principal Investigator — Assistant Professor, Jazan University
Locations (1):
- Jazan University, Jizan, Gizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmed MM, Alawna M, Youssef ASA, Amin WM, Alajam RA, Morsy WE, Fayed E, Mohamed AA. Immediate effect of physical activity on the autonomic nervous system in individuals with autism spectrum disorders of different age groups: a randomised trial. BMJ Open Sport Exerc Med. 2024 Apr 11;10(2):e001822. doi: 10.1136/bmjsem-2023-001822. eCollection 2024. PMID 38617566